CLINICAL TRIAL: NCT04682561
Title: The STEP Program: Building Trauma Resilience Among Nurses and Personal Support Workers Across Ontario During and Beyond the COVID-19 Pandemic
Brief Title: STEP: Building Trauma Resilience Among Nurses and Personal Support Workers During and Beyond COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Providence Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP-01
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-08

CONDITIONS: Stress; Trauma; Mental Health Issue; Healthcare Workers
Keywords: Stress Prevention; Trauma Coping; Psychotherapy; COVID-19; Nurse; Personal Support Worker
MeSH Terms: conditions — Wounds and Injuries; COVID-19

STUDY DESIGN:
Intervention Model Description: 3 month, within-subjects longitudinal study, with each participant receiving 8 weekly sessions of the STEP psychotherapy intervention designed to help mitigate the effects of stress and trauma on their ability to provide patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Trauma Exposure Preparation (STEP) Program (Experimental): Nurses or personal support workers in Ontario will undergo the STEP Program Psychotherapy
  Interventions: Behavioral: Supportive Trauma Exposure Preparation Program

INTERVENTIONS:
Behavioral: Supportive Trauma Exposure Preparation Program — The Supportive Trauma Exposure Preparation Program is based on the theory that the ability to set compassionate boundaries will enhance acceptance of the reality of trauma in the workplace, and will also increase the cognitive/emotional/physical energy needed to engage in adaptive emotional strategies in response to trauma exposure. Therefore, the goal of therapy is to learn to set compassionate boundaries and engage with oneself and others from a perspective of self-empowerment and acceptance of life events. Concepts and skills will be addressed through the following modules: 1) understanding of trauma and its effects, 2) personal rights and boundaries, 3) emotional literacy, 4) distress tolerance and emotion regulation skills building, 5) communication skills building, 6) self-compassion and acceptance, and 7) enhancing self-care.
  Other Names: STEP Program

SUMMARY:
The COVID-19 pandemic has amplified the need for skills training and mental health support for healthcare workers who are exposed to the numerous stressors and potential trauma of a high-risk environment. This context is associated with significant impacts on mental health, including depression, anxiety, and post-traumatic stress, with nurses and personal support workers (PSWs) being disproportionately impacted. The proposed STEP program is an intervention that aims to equip nurses and PSWs with the skills and support needed to promote their wellness and navigate the challenges of experiencing trauma in a high-risk, high-stress environment, which has been exacerbated by the pandemic. As such, the STEP intervention has the potential to improve trauma resilience and mental health among nurses and PSW, which may ultimately improve patient care and benefit the hospital system during and even beyond the pandemic. The results from this study will also provide vital insight into promising interventions for healthcare workers that are accessible and scalable.

DETAILED DESCRIPTION:
Conducting work where exposure to trauma occurs requires specific resources and skillsets to manage the immense mental and emotional side effects that can arise. Notably, some nurses and personal support workers (PSWs) deal with trauma on a regular basis, yet often do not have access to such training. It is not surprising, then, that estimates of compassion fatigue and burnout are a staggering 40-60% among healthcare workers, This has been shown to have direct negative effects on personal wellness, patient care, workplace functioning, and the hospital system. Factors that contribute to compassion fatigue include being exposed to another's suffering and stressful work environments. Notably, the COVID-19 pandemic has exacerbated these factors. Furthermore, reduced staffing, increased exposure to trauma, and enhanced perceptions of workplace threat during a pandemic are additional factors that have been shown to significantly impact the mental health and wellness of frontline workers. The need for adequate supports for these frontline workers is essential during and beyond the COVID-19 pandemic. The vast majority of workplace-based organizational interventions for mental health concerns among healthcare workers are delivered in a group setting, primarily focused on psychoeducation and stress reduction techniques.Very few programs include a component involving one-on-one psychotherapy with a licensed therapist, and when offered, it is typically an event-triggered counselling session (i.e., a therapist is made available to a participant in the case where they experience a traumatic stressor at work, such as a bereavement case or managing a patient with traumatic injury. Numerous editorials have been published since the start of the pandemic calling for mental health support for healthcare workers. Among the supportive measures that have been consistently recommended in these reports are the following: provide education on stress and mental health to validate experience; offer stress management, resilience and coping skills training; incorporate debriefing practices; facilitate morale boosting; and offer psychological support through a licensed therapist. We have developed the Supportive Trauma Exposure Preparation (STEP) program to address these unmet critical needs and suggested recommendations. The STEP program is an 8-week psychotherapy intervention designed to teach concepts, skills and coping strategies to healthcare workers with the aim of improving mental health and building resilience in the face of trauma/stress exposure in the healthcare workplace setting. This is a pilot study exploring the effectiveness and feasibility/acceptability of the STEP intervention in reducing burnout, building resilience and improving mental health outcomes for nurses and personal support workers in Ontario. The STEP program has the potential to be widely accessible and fit the demanding work schedule of healthcare workers. Such a program would be useful even beyond the pandemic, given the nature of the healthcare providers' work and what is known about the high prevalence and consequences of stress and compassion fatigue in the pre-COVID-19 pandemic context.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a nurse or personal support worker in Ontario
* 18 years or older
* Access to a computer with a camera or a mobile phone with a camera
* Access to internet
* Not receiving other psychotherapy concurrently
* Follow-up visits with a psychiatrist or family doctor where a psychotherapeutic modality (e.g. cognitive-behavioural therapy, etc.) is not being used are allowable.
* Able to undergo psychotherapy in English
* Working a minimum of 1 shift per week in a hospital setting or community long term care home

Exclusion Criteria:

* Unable to commit to 1-hour weekly psychotherapy session for the 8 weeks duration of the study
* Individuals with current high risk for suicide, alcohol or substance use, or active psychosis at the time of screening will not be eligible. Recommendations will be made to appropriate mental health services (e.g., Employee Assistance Program, physician referral to psychiatrist, Ontario COVID-19 Mental Health Network) in order to connect the individual to more targeted support and intervention.
* The presence of cognitive impairment (based on clinical judgment) that would limit consent or understanding of STEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to post-intervention in healthcare worker burnout using Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL) burnout subscale | Baseline, week 4, week 8 and 3 months
  The ProQOL is a 30-item self-report questionnaire assessing negative and positive effects of helping others who experience suffering and trauma, with subscales for compassion satisfaction, burnout and compassion fatigue. Focus will be paid to the burnout subscale score.

SECONDARY OUTCOMES:
Changes in healthcare worker resilience using Connor-Davidson Resilience Scale 10 item (CD-RISC 10) | Baseline, week 8, and 3 months
  The CD-RISC 10 is a 10-item self-report scale used to measure ability to cope with stress and adversity as an indicator of resilience.
Changes in healthcare worker depression symptoms using Patient Health Questionnaire - 9 item (PHQ-9) | Baseline, weeks 2-8, and 3 months
  The PHQ-9 is a 9-item self-report scale assessing depression symptoms.Total scores range from 0 to 27, with higher scores reflecting more severe anxiety. Focus will be paid to changes in depression symptom severity.
Changes in healthcare worker anxiety symptoms using Generalized Anxiety Disorder 7-item scale (GAD-7) | Baseline, weeks 2-8, and 3 months
  The GAD-7 is a brief 7-item self-report scale measuring anxiety symptoms. Total scores range from 0 to 21, with higher scores reflecting more severe anxiety. Focus will be paid to changes in anxiety severity.
Changes in healthcare worker compassion satisfaction and secondary traumatic stress subscales of the Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL) | Baseline, week 4, week 8 and 3 months
  The ProQOL is a 30-item self-report questionnaire assessing negative and positive effects of helping others who experience suffering and trauma, with subscales for compassion satisfaction, burnout and compassion fatigue.
Changes in healthcare worker perceived quality of patient care | Baseline, weeks 2-8, and 3 months
  This will be assessed by asking participants to rate their perception of the quality of patient care they provided on their last shift, using a 4-point Likert scale.
Changes in Sheehan Disability Scale (SDS) score | Baseline, week 4, week 8, and 3 months
  The SDS is a brief 3-item self-report scale that probes work/school, social, and family/home functioning. Each item is scored from 0 to 10. Total scores range from 0 (unimpaired) to 30 (highly impaired).
Changes in The Lam Employment Absence and Productivity Scale (LEAPS) score | Baseline, week 2, week 4, week 6, week 8 and 3 months
  The LEAPS is a 10-item, self-rated scale that provides a measure of functioning at work.

OTHER OUTCOMES:
Participant feedback on their experiences with specific aspects of the STEP program | 3 months
  Feasibility and Acceptability survey and interview created in-house with questions designed to collect quantitative and qualitative feedback from participants with respect to the feasibility and acceptability of the STEP Program

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lalovic A, Hyde M, Bergmans Y, Kiriakidis A, Ebegbare N, Verduyn A, Rizvi SJ. Enhancing Trauma Resilience in Nurses and Personal Support Workers: A Feasibility Study of an 8-Week Supportive Trauma Exposure Preparation Intervention. Can J Nurs Res. 2025 Dec;57(4):580-591. doi: 10.1177/08445621251354918. Epub 2025 Jun 30. PMID 40589165